CLINICAL TRIAL: NCT00515190
Title: A Randomized Phase II Study of Continuous or Intermittent S-1 Combined With Oxaliplatin in Recurrent or Metastatic Gastric Carcinoma
Brief Title: Study of Continuous or Intermittent S-1 Combined With Oxaliplatin in Recurrent or Metastatic Gastric Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Sook Ryun Park, M.D., National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-265; 82-31-920-1609
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Secondary; Combination chemotherapy; S-1; oxaliplatin
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): (continuous):S-1 plus oxalipatin will be continued until disease progression, unacceptable toxicity or consent withdrawal.
  Interventions: Drug: S-1,oxaliplatin
- B (Active Comparator): (intermittent arm): Treatment will be stopped after the initial 6 cycles of S-1 plus oxaliplatin, and then S-1 plus oxaliplatin will be resumed at the disease progression during follow-up, as the same dose as the last chemotherapy of initial 6 cycles.
  Interventions: Drug: S-1,oxaliplatin

INTERVENTIONS:
Drug: S-1,oxaliplatin — Arm A (continuous arm): S-1 80mg/m2/d p.o. twice daily(q 12-h)on D1(evening)-D15(morning)plus oxaliplatin 130mg/m2 IV(in the vein)on D1 every 3 weeks, until disease progression, unacceptable toxicity, or consent withdrawal.
  Arm B (intermittent arm):Treatment will be stopped after the initial 6 cycles of S-1 plus oxaliplatin, and then S-1 plus oxaliplatin will be resumed at the disease progression during follow-up, as the same dose as the last chemotherapy of initial 6 cycles.

SUMMARY:
Randomized phase II study designed to evaluate the efficacy and safety of continuous S-1 plus oxaliplatin versus intermittent S-1 plus oxaliplatin as first-line therapy in patients with recurrent and/or metastastic gastric carcinoma. Within 2 weeks of the end of induction chemotherapy of 6 cycles with S-1 plus oxalipatin, patients who don't experience progression will be randomized to the continuous S-1 plus oxaliplatin arm or the intermittent S-1 plus oxaliplatin arm in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed gastric adenocarcinoma with recurrent and/or metastatic disease
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) or non-measurable evaluable
5. No prior treatment for recurrent and/or metastatic disease (prior adjuvant/neoadjuvant therapy is allowed if at least 6 months has elapsed between completion of adjuvant/neoadjuvant therapy and enrolment into the study; prior oxaliplatin is not allowed)
6. Adequate major organ function including the following: Hematopoietic function: ANC >= 1,500/mm3, Platelet >= 100,000/mm3, Hepatic function: serum bilirubin =< 1.5 x ULN, AST/ALT levels =< 2.5 x ULN (=< 5 x ULN if liver metastases are present)Renal function: serum creatinine =< 1.5 x ULN
7. Patients should sign a written informed consent before study entry

Exclusion Criteria:

1. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome (e.g. patients with partial or total gastrectomy can enter the study, but not those with a jejunostomy probe), or inability to take oral medication
2. Patients with active (significant or uncontrolled) gastrointestinal bleeding
3. Residual relevant toxicity resulting from previous therapy (with the exception of alopecia) ≥ grade 2 NCI-CTCAE version 3.0
4. Prior and/or current history of peripheral neuropathy

   * grade 1 NCI-CTCAE version 3.0
5. Inadequate cardiovascular function:New York Heart Association class III or IV heart diseaseUnstable angina or myocardial infarction within the past 6 monthsHistory of significant ventricular arrhythmia requiring medication with antiarrhythmics or significant conduction system abnormality
6. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy
7. Other malignancy within the past 3 years except non-melanomatous skin cancer or carcinoma in situ of the cervix
8. History of or current brain metastases
9. Psychiatric disorder that would preclude compliance
10. Females with a positive or no pregnancy test (within 7 days before treatment start) until childbearing potential can be otherwise excluded (postmenopausal i.e. amenorrheic for at least 2 years, hysterectomy or oophorectomy)
11. Subjects with reproductive potential not willing to use an effective method of contraception
12. Lactating women
13. Known dihydropyrimidine dehydrogenase deficiency
14. Patients receiving a concomitant treatment with drugs interacting with S-1 such as flucytosine, phenytoin, or warfarin et al.
15. Major surgery within 4 weeks of start of study treatment, without complete recovery
16. Radiotherapy within 4 weeks of start of study treatment; 2 weeks interval allowed if palliative radiotherapy was given to bone metastatic site and patient recovered from any acute toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2007-07; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Overall survial in the two treatment arms | During study period

SECONDARY OUTCOMES:
Response rate, toxicity, duration of response, time to progression, Quality of life in the two treatment arms,the effect of CYP2A6 genetic polymorphisms on the pharmacokinetics, treatment efficacy and toxicity | During study period

CONTACTS AND LOCATIONS:
Overall Officials: Sook Ryun Park, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea